CLINICAL TRIAL: NCT01262118
Title: An Exploratory Phase 1, Fixed Sequence, Open-Label Study To Assess The Effects Of CP-690,550 On The Kinetics Of Cholesterol Flux Through The High Density Lipoprotein/Reverse Cholesterol Transport Pathway In Patients With Active Rheumatoid Arthritis
Brief Title: Effects Of CP-690,550 (Tasocitinib) On Cholesterol Metabolism In Patients With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A3921130
Record Dates: First submitted 2010-11-15; First posted 2010-12-17 (Estimated); Results first posted 2013-01-23 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2012-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Cholesterol metabolism; Cholesterol flux; Rheumatoid Arthritis; Tasocitinib; CP-690; 550
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CP-690,550 (tasocitinib) 10 mg twice daily (BID) (Experimental)
  Interventions: Drug: CP-690,550 (tasocitinib)
- Healthy Volunteers (No Intervention): No intervention

INTERVENTIONS:
Drug: CP-690,550 (tasocitinib) — CP-690,550 (tasocitinib) dosed at 10 mg BID for 6 weeks in patients with active rheumatoid arthritis
  Arms: CP-690,550 (tasocitinib) 10 mg twice daily (BID)

SUMMARY:
The purpose of study is to explore the effect of CP-690,550 (tasocitinib) on cholesterol metabolism in patients with active rheumatoid arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

* Males or females, 18 years of age or older with active rheumatoid arthritis; Or male and female healthy volunteers 18 years of age and older

Exclusion Criteria:

* Pregnant or lactating women
* Clinically significant systemic disease (other than RA for RA arm)
* Use of lipid-regulating agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2011-05; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- United States (8):
  - Pfizer Investigational Site, Anniston, Alabama
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Daytona Beach, Florida
  - Pfizer Investigational Site, Ormond Beach, Florida
  - Pfizer Investigational Site, South Miami, Florida
  - Pfizer Investigational Site, Bingham Farms, Michigan
  - Pfizer Investigational Site, Dallas, Texas
- Hungary (2):
  - Pfizer Investigational Site, Balatonfüred
  - Pfizer Investigational Site, Budapest

REFERENCES:
- [Derived] Kristensen LE, Danese S, Yndestad A, Wang C, Nagy E, Modesto I, Rivas J, Benda B. Identification of two tofacitinib subpopulations with different relative risk versus TNF inhibitors: an analysis of the open label, randomised controlled study ORAL Surveillance. Ann Rheum Dis. 2023 Jul;82(7):901-910. doi: 10.1136/ard-2022-223715. Epub 2023 Mar 17. PMID 36931693
- [Derived] Hansen KE, Mortezavi M, Nagy E, Wang C, Connell CA, Radi Z, Litman HJ, Adami G, Rossini M. Fracture in clinical studies of tofacitinib in rheumatoid arthritis. Ther Adv Musculoskelet Dis. 2022 Dec 27;14:1759720X221142346. doi: 10.1177/1759720X221142346. eCollection 2022. PMID 36601090
- [Derived] Curtis JR, Yamaoka K, Chen YH, Bhatt DL, Gunay LM, Sugiyama N, Connell CA, Wang C, Wu J, Menon S, Vranic I, Gomez-Reino JJ. Malignancy risk with tofacitinib versus TNF inhibitors in rheumatoid arthritis: results from the open-label, randomised controlled ORAL Surveillance trial. Ann Rheum Dis. 2023 Mar;82(3):331-343. doi: 10.1136/ard-2022-222543. Epub 2022 Dec 5. PMID 36600185
- [Derived] Winthrop KL, Yndestad A, Henrohn D, Danese S, Marsal S, Galindo M, Woolcott JC, Jo H, Kwok K, Shapiro AB, Jones TV, Diehl A, Su C, Panes J, Cohen SB. Influenza Adverse Events in Patients with Rheumatoid Arthritis, Ulcerative Colitis, or Psoriatic Arthritis in the Tofacitinib Clinical Development Programs. Rheumatol Ther. 2023 Apr;10(2):357-373. doi: 10.1007/s40744-022-00507-z. Epub 2022 Dec 17. PMID 36526796
- [Derived] Winthrop KL, Curtis JR, Yamaoka K, Lee EB, Hirose T, Rivas JL, Kwok K, Burmester GR. Clinical Management of Herpes Zoster in Patients With Rheumatoid Arthritis or Psoriatic Arthritis Receiving Tofacitinib Treatment. Rheumatol Ther. 2022 Feb;9(1):243-263. doi: 10.1007/s40744-021-00390-0. Epub 2021 Dec 6. PMID 34870800
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Wang L, Chen C, Kwok K, Biswas P, Shapiro A, Madsen A, Wollenhaupt J. Long-term safety of tofacitinib up to 9.5 years: a comprehensive integrated analysis of the rheumatoid arthritis clinical development programme. RMD Open. 2020 Oct;6(3):e001395. doi: 10.1136/rmdopen-2020-001395. PMID 33127856
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Thirunavukkarasu K, DeMasi R, Geier J, Kwok K, Wang L, Riese R, Wollenhaupt J. Long-term safety of tofacitinib for the treatment of rheumatoid arthritis up to 8.5 years: integrated analysis of data from the global clinical trials. Ann Rheum Dis. 2017 Jul;76(7):1253-1262. doi: 10.1136/annrheumdis-2016-210457. Epub 2017 Jan 31. PMID 28143815
- [Derived] Charles-Schoeman C, Fleischmann R, Davignon J, Schwartz H, Turner SM, Beysen C, Milad M, Hellerstein MK, Luo Z, Kaplan IV, Riese R, Zuckerman A, McInnes IB. Potential mechanisms leading to the abnormal lipid profile in patients with rheumatoid arthritis versus healthy volunteers and reversal by tofacitinib. Arthritis Rheumatol. 2015 Mar;67(3):616-25. doi: 10.1002/art.38974. PMID 25470338
- [Derived] Cohen S, Radominski SC, Gomez-Reino JJ, Wang L, Krishnaswami S, Wood SP, Soma K, Nduaka CI, Kwok K, Valdez H, Benda B, Riese R. Analysis of infections and all-cause mortality in phase II, phase III, and long-term extension studies of tofacitinib in patients with rheumatoid arthritis. Arthritis Rheumatol. 2014 Nov;66(11):2924-37. doi: 10.1002/art.38779. PMID 25047021
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921130&StudyName=Effects%20Of%20CP-690%2C550%20%28Tasocitinib%29%20On%20Cholesterol%20Metabolism%20In%20Patients%20With%20Active%20Rheumatoid%20Arthritis%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Rheumatoid Arthritis Cohort: Active rheumatoid arthritis participants were assessed for baseline cholesterol flux kinetics for 3 days and then received CP-690,550 10 mg tablet orally twice daily for 6 weeks.
- Healthy Volunteers Cohort: Healthy volunteers with similar baseline demographic characteristics as the active rheumatoid arthritis participants were assessed for baseline cholesterol flux kinetics for 3 days.
Period: Baseline Assessment Period (3 Days)
Arm/Group | Rheumatoid Arthritis Cohort | Healthy Volunteers Cohort
Started | 36 | 33
Completed | 36 | 33
Not Completed | 0 | 0
Period: Treatment Period (6 Weeks)
Arm/Group | Rheumatoid Arthritis Cohort | Healthy Volunteers Cohort
Started | 36 | 0
Completed | 36 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rheumatoid Arthritis Cohort | Healthy Volunteers Cohort | Total
Number analyzed (Participants) | 36 | 33 | 69
Age, Customized [Number; unit: participants]
  18 to 44 years | 9 | 7 | 16
  45 to 64 years | 25 | 25 | 50
  Greater than or equal to (>=) 65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 28 | 58
  Male | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: High-density Lipoprotein Cholesterol (HDL-C) Concentration at Baseline
Description: Blood level of HDL-C was measured following a 12-hours fasting.
Time Frame: Baseline
Population: Full analysis set (FAS) included all enrolled participants who had any measurement of cholesterol ester production rate available.
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Groups:
- Healthy Volunteer Cohort: Healthy volunteers with similar baseline demographic characteristics as the active rheumatoid arthritis participants were assessed for baseline cholesterol flux kinetics for 3 days.
Arm/Group | Rheumatoid Arthritis Cohort | Healthy Volunteer Cohort
Number analyzed (Participants) | 36 | 31
milligram per deciliter (mg/dL) | 54.30 (12.52) | 63.43 (16.89)

2. Primary Outcome: High-density Lipoprotein Cholesterol (HDL-C) Concentration at Week 6
Description: Blood level of HDL-C was measured following a 12-hours fasting.
Time Frame: Week 6
Population: FAS included all enrolled participants who had any measurement of cholesterol ester production rate available.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Rheumatoid Arthritis Cohort
Number analyzed (Participants) | 36
mg/dL | 62.34 (15.24)

3. Primary Outcome: Cholesterol Ester Production Rate at Baseline
Description: Cholesterol ester production rate was calculated using a 3-pool model with a simulation, analysis and modeling (SAAM II) program.
Time Frame: Baseline
Population: FAS included all enrolled participants who had any measurement of cholesterol ester production rate available. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: (mg per kilogram) per hour ([mg/kg]/hr)
Arm/Group | Rheumatoid Arthritis Cohort | Healthy Volunteer Cohort
Number analyzed (Participants) | 34 | 31
(mg per kilogram) per hour ([mg/kg]/hr) | 1.09 (0.24) | 1.11 (0.26)

4. Primary Outcome: Cholesterol Ester Production Rate at Week 6
Description: as for outcome 3
Time Frame: Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: (mg/kg)/hr
Arm/Group | Rheumatoid Arthritis Cohort
Number analyzed (Participants) | 33
(mg/kg)/hr | 1.12 (0.24)

5. Secondary Outcome: Low-density Lipoprotein Cholesterol (LDL-C) and Total Cholesterol Concentration
Description: Blood level of LDL-C and total cholesterol (TC) was measured following a 12-hours fasting.
Time Frame: Baseline, Week 6
Population: FAS included all enrolled participants who had any measurement of cholesterol ester production rate available.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Rheumatoid Arthritis Cohort | Healthy Volunteer Cohort
Number analyzed (Participants) | 36 | 31
mg/dL
  Baseline: LDL-C | 124.61 (28.55) | 144.88 (36.36)
  Baseline: TC | 193.79 (32.56) | 221.57 (42.12)
  Week 6: LDL-C | 142.68 (39.02) | NA (NA) — Data not available at this time point since as per analysis plan healthy volunteers were enrolled only for baseline assessment period.
  Week 6: TC | 219.83 (41.33) | NA (NA) — Data not available at this time point since as per analysis plan healthy volunteers were enrolled only for baseline assessment period.

6. Secondary Outcome: Cholesterol Ester Fractional Catabolic Rate
Description: Cholesterol ester fractional catabolic rate were calculated using a 3-pool model with a simulation, analysis and modeling (SAAM II) program. Fractional catabolic rate was the percentage of cholesterol ester which was replaced, transferred or lost per unit of time.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage ester per hour (%/hr)
Arm/Group | Rheumatoid Arthritis Cohort | Healthy Volunteer Cohort
Number analyzed (Participants) | 34 | 31
percentage ester per hour (%/hr)
  Baseline | 2.43 (0.39) | 2.17 (0.36)
  Week 6 | 2.23 (0.31) | NA (NA) — Data not available at this time point since as per analysis plan healthy volunteers were enrolled only for baseline assessment period.

7. Secondary Outcome: Low-density Lipoprotein Associated With Apolipoprotein B (LDL-apoB) Production Rate
Description: LDL-apoB production rate were calculated using a 3-pool model with a simulation, analysis and modeling (SAAM II) program.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: (mg/kg)/hr
Arm/Group | Rheumatoid Arthritis Cohort | Healthy Volunteer Cohort
Number analyzed (Participants) | 32 | 30
(mg/kg)/hr
  Baseline | 0.49 (0.12) | 0.50 (0.13)
  Week 6 | 0.52 (0.12) | NA (NA) — Data not available at this time point since as per analysis plan healthy volunteers were enrolled only for baseline assessment period.

8. Secondary Outcome: Low-density Lipoprotein Associated With Apolipoprotein B (LDL-apoB) Fractional Catabolic Rate
Description: Fractional catabolic rate for LDL ApoB were calculated using the 13 carbon (13C) isotopic enrichment of very low density lipoprotein (VLDL) as the limiting value. Isotope 13C in plasma was measured using Gas Chromatography-Combustion-Isotope Ratio Mass Spectrometry (GC-C-IRMS).
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: %/hr
Arm/Group | Rheumatoid Arthritis Cohort | Healthy Volunteer Cohort
Number analyzed (Participants) | 32 | 30
%/hr
  Baseline | 1.61 (0.37) | 1.50 (0.35)
  Week 6 | 1.57 (0.41) | NA (NA) — Data not available at this time point since as per analysis plan healthy volunteers were enrolled only for baseline assessment period.

9. Secondary Outcome: High-density Lipoprotein Associated With Apolipoprotein A1 (HDL-apoA1) Production Rate
Description: HDL-apoA1 production rate were calculated using a 3-pool model with a simulation, analysis and modeling (SAAM II) program.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/kg/hr
Arm/Group | Rheumatoid Arthritis Cohort | Healthy Volunteer Cohort
Number analyzed (Participants) | 32 | 30
mg/kg/hr
  Baseline | 0.57 (0.11) | 0.59 (0.16)
  Week 6 | 0.65 (0.15) | NA (NA) — Data not available at this time point since as per analysis plan healthy volunteers were enrolled only for baseline assessment period.

10. Secondary Outcome: High-density Lipoprotein Associated With Apolipoprotein A1 (HDL-apoA1) Fractional Catabolic Rate
Description: Fractional catabolic rate for HDL-apoA1 were calculated using the 13C isotopic enrichment of VLDL as the limiting value. Isotope 13C in plasma was measured using GC-C-IRMS.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: %/hr
Arm/Group | Rheumatoid Arthritis Cohort | Healthy Volunteer Cohort
Number analyzed (Participants) | 32 | 30
%/hr
  Baseline | 1.08 (0.22) | 1.02 (0.22)
  Week 6 | 1.11 (0.28) | NA (NA) — Data not available at this time point since as per analysis plan healthy volunteers were enrolled only for baseline assessment period.

11. Secondary Outcome: Cholesterol Efflux Rate
Description: Cholesterol efflux rate was measured using isotope dilution method in which rate of appearance of isotope 13C-free cholesterol in plasma representing whole body efflux from tissues was assessed. Isotope 13C in plasma was measured using GC-C-IRMS.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: (mg/kg)/hr
Arm/Group | Rheumatoid Arthritis Cohort | Healthy Volunteer Cohort
Number analyzed (Participants) | 34 | 31
(mg/kg)/hr
  Baseline | 4.02 (0.96) | 4.35 (1.53)
  Week 6 | 4.04 (1.08) | NA (NA) — Data not available at this time point since as per analysis plan healthy volunteers were enrolled only for baseline assessment period.

ADVERSE EVENTS:
Arm/Group | Rheumatoid Arthritis Cohort | Healthy Volunteer Cohort
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/33
Other Adverse Events (participants affected / at risk) | 19/36 | 6/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rheumatoid Arthritis Cohort (N=36) | Healthy Volunteer Cohort (N=33)
Abdominal distension (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Irritability (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 1
Sinusitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 7 | 0
Urinary tract infection (Infections and infestations) | 3 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 4 | 4
Migraine (Nervous system disorders) | 1 | 1
Sciatica (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.